CLINICAL TRIAL: NCT00941057
Title: Open-label, Randomized, Cross-over Study to Investigate the Bioequivalence of Estradiol Valerate (EV), Dienogest (DNG) and Levomefolate Calcium After Single Oral Administration of a Tablet Formulation Containing 2 mg Estradiol Valerate and 3 mg Dienogest Without and With 0.451 mg Levomefolate Calcium and a Tablet Formulation Containing 0.451 mg Levomefolate Calcium in 42 Healthy Postmenopausal Women
Brief Title: Bioequivalence Study: 2 mg Estradiol Valerate (EV) and 3 mg Dienogest (DNG) Without and With Levomefolate Calcium
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: 13469; 2009-011963-35 (EudraCT Number)
Record Dates: First submitted 2009-07-16; First posted 2009-07-17 (Estimated); Last update posted 2016-08-01 (Estimated); Status verified 2016-07

CONDITIONS: Pharmacology, Clinical
MeSH Terms: interventions — dienogest; levomefolate calcium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Estradiol + dienogest + levomefolate (Experimental): Treatment A
  Interventions: Drug: BAY 98-7079, Estradiolvalerate (EV) / Dienogest (DNG) / Levomefolate calcium
- Estradiol + dienogest (Active Comparator): Treatment B
  Interventions: Drug: BAY 86-5027,Estradiolvalerate(EV) / Dienogest (DNG)
- Levomefolate (Active Comparator): Treatment C
  Interventions: Drug: BAY 86-7660,levomefolate calcium

INTERVENTIONS:
Drug: BAY 98-7079, Estradiolvalerate (EV) / Dienogest (DNG) / Levomefolate calcium — Oral, single dose, 2 mg EV + 3 mg DNG + 0.451 mg levomefolate calcium washout phase between treatments: at least 7 days
  Arms: Estradiol + dienogest + levomefolate
Drug: BAY 86-5027,Estradiolvalerate(EV) / Dienogest (DNG) — Oral, single dose, 2 mg EV + 3 mg DNG washout phase between treatments: at least 7 days
  Arms: Estradiol + dienogest
Drug: BAY 86-7660,levomefolate calcium — Oral, single dose, 0.451 mg levomefolate calcium washout phase between treatments: at least 7 days
  Arms: Levomefolate

SUMMARY:
Investigation of the bioequivalence (BE) of Estradiol Valerate (EV) and Dienogest (DNG) after administration of one film-coated tablet containing 2 mg Estradiol Valerate, 3 mg Dienogest and 0.451 mg Levomefolate calcium as compared to one film-coated tablet containing 2 mg Estradiol Valerate,3 mg Dienogest.Investigation of the bioequivalence of levomefolate calcium after administration of one film-coated tablet containing 2 mg Estradiol Valerate, 3 mg Dienogest and 0.451 mg Levomefolate calcium as compared to one film-coated tablet containing 0.451 mg levomefolate calcium

ELIGIBILITY:
Inclusion Criteria:

* Healthy postmenopausal women, age: 45-75 years with body mass index between ≥18 and ≤30 kg/m2. Post-menopausal state revealed by: medical history, and hormone analyses in serum: estradiol ≤20 pg/mL and in women <60 years old: follicle-stimulating hormone ≥ 40 IU/L at screening

Exclusion Criteria:

* Contraindications for use of combined (Estradiolvalerate/Dienogest) contraceptive (e.g.history of venous/arterial thromboembolic disease)
* Regular intake of medication
* Clinically relevant findings (ECG, blood pressure, physical and gynaecological examination, laboratory examination)
* Smoking

Ages: 45 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2009-09; Primary Completion 2009-12 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
AUC | Pre-dose and up to 72 hr post-dose for the treatments A and B and up to 12 hr post dose for the treatment C
  Area under the concentration vs time curve from zero to infinity for DNG
Cmax | Pre-dose and up to 72 hr post-dose for the treatments A and B and up to 12 hr post dose for the treatment C
  Maximum drug concentration for DNG and for E1, E2, E1S, and L-5-methyl-THF (baseline corrected and uncorrected)
AUC(0-tlast) | Pre-dose and up to 72 hr post-dose for the treatments A and B and up to 12 hr post dose for the treatment C
  AUC from time 0 to the last data point above the lower limit of quantitation for E1, E2, E1S, and L-5-methyl-THF (baseline corrected and uncorrected)

SECONDARY OUTCOMES:
tmax | Pre-dose and up to 72 hr post-dose for the treatments A and B and up to 12 hr post dose for the treatment C
  Time to reach maximum drug concentration in plasma for DNG and E1, E2, E1S, and L-5-methyl-THF (baseline uncorrected)
t½ | Pre-dose and up to 72 hr post-dose for the treatments A and B and up to 12 hr post dose for the treatment C
  Half-life associated with the terminal slope for DNG and E1, E2, E1S, and L-5-methyl-THF
λz | Pre-dose and up to 72 hr post-dose for the treatments A and B and up to 12 hr post dose for the treatment C
  Apparent terminal rate constant(estimates only) for DNG and E1, E2, E1S, and L-5-methyl-THF
AUC(0-tlast) | Pre-dose and up to 72 hr post-dose for the treatments A and B and up to 12 hr post dose for the treatment C
  AUC from time 0 to the last data point above the lower limit of quantitation for DNG
AUC | Pre-dose and up to 72 hr post-dose for the treatments A and B and up to 12 hr post dose for the treatment C
  Area under the concentration vs time curve from zero to infinity E1, E2, E1S, and L-5-methyl-THF (baseline corrected)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Neu-Ulm, Bavaria, Germany

REFERENCES:
- See also: Click here to find information about studies related to Bayer Healthcare products conducted in Europe. — http://www.clinicaltrialsregister.eu/